CLINICAL TRIAL: NCT06241703
Title: Effect of Intermittent Urethral Catheter Clamping Combined With Active Urination Training (ICCAUT) Strategy on Postoperative Urinary Dysfunction After Radical Rectal Cancer Surgery: a Single-Center Randomized Controlled Trial (ICCAUT-1)
Brief Title: Effect of ICCAUT Strategy on Postoperative Urinary Dysfunction After Radical Rectal Cancer Surgery
Acronym: ICCAUT-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yuchen Guo, Ph.D., Prof., The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICCAUT-1
Record Dates: First submitted 2024-01-17; First posted 2024-02-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Urinary Dysfunction; Rectal Cancer; Urinary Catheterization; Urinary Retention Postoperative
Keywords: Residual Urine Volume; Urinary Retention; Urinary Dysfunction; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms; Urinary Retention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patients and bedside nurses cannot be blinded, but the attending physicians and the medical ultrasound doctor will be blinded. The medical team will ensure that the patients and bedside nurses keep the group assignment confidential from the attending physicians and the medical ultrasound doctor. Unblinding will occur when the patient is discharged, and any instances of premature unblinding will be recorded. Additionally, the data analysts involved in this study will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICCAUT Group (Experimental): Patients undergoing laparoscopic/robotic rectal cancer TME surgery will undergo bladder training. The bladder training include intermittent catheter clamping and active urination to facilitate complete bladder emptying each time the catheter is released, which we called ICCAUT strategy. The training will commence at 9:00 am on the first postoperative day, and the catheter will be removed at 9:00 am on the second postoperative day after the bladder is empty.
  Interventions: Procedure: ICCAUT
- Free Drainage Group (Other): Patients undergoing laparoscopic/robotic rectal cancer TME surgery will have their urinary catheter kept open postoperatively, and the catheter will be removed at 9:00 am on the second postoperative day.
  Interventions: Procedure: Free drainage

INTERVENTIONS:
Procedure: ICCAUT — For patients in the ICCAUT group, intermittent catheter clamping will be initiated at 9:00 AM. The catheter will be clamped for 3 h, followed by a 5-minute release, which is one cycle. The next cycle will begin after the cycle was completed. Catheter training is to conclude at 10:00 PM on the first postoperative day, and the catheter is left open during the night. At 6:00 AM on the second postoperative day, another cycle of catheter training will be performed, with the catheter removed at 9:00 AM after the bladder is empty. During the training period, if the patient experiences a strong urge to urinate before the 3-hour clamping time is over, the clamping can be released in advance for 5 min, allowing the patient to proceed to the next cycle of bladder training. Each time the catheter is released, we will encourage the patients to actively initiate urination to facilitate complete bladder emptying.
  Arms: ICCAUT Group
Procedure: Free drainage — For patients in the free draining group, no intervention will be performed on the catheter during this period. The catheter will be removed at 9:00 AM on postoperative day two.
  Arms: Free Drainage Group

SUMMARY:
In this study, the bladder training include intermittent urethral catheter clamping combined with active urination training, which the investigators called ICCAUT strategy. This prospective, single-center, randomized controlled trial will recruit participants with rectal cancer. The participants will be randomly assigned in a 1:1 ratio to either the ICCAUT group or the free-drainage group. In the ICCAUT group, the participants will undergo intermittent clamping of the urinary catheter prior to its removal. Each time the catheter is released, the investigators will encourage the participants to actively initiate urination to facilitate complete bladder emptying. While participants in the free-drainage group will not receive any specific training. The urinary catheter will be removed on the second day after the surgery for both groups after the bladder is empty. The primary endpoint is the incidence of urinary dysfunction, which include secondary catheterization or incomplete bladder emptying. Secondary endpoints include urinary tract infection, time to first urination after catheter removal, catheter-related bladder discomfort syndrome, postoperative morbidity and mortality, as well as urinary function within 30 days.

DETAILED DESCRIPTION:
Urinary catheter placement is a routine procedure performed in proctectomy. Nevertheless, there is uncertainty regarding the need for bladder training before catheter removal. The purpose of this trial is to examine the impact of bladder training on the urinary retention and secondary catheterization following proctectomy.

In this study, the bladder training include intermittent urethral catheter clamping combined with active urination training, which the investigators called ICCAUT strategy. This prospective, single-center, randomized controlled trial will recruit participants with rectal cancer. The participants will be randomly assigned in a 1:1 ratio to either the ICCAUT group or the free-drainage group. In the ICCAUT group, the participants will undergo intermittent clamping of the urinary catheter prior to its removal. Each time the catheter is released, the investigators will encourage the participants to actively initiate urination to facilitate complete bladder emptying. While the participants in the free-drainage group will not receive any specific training. The urinary catheter will be removed on the second day after the surgery for both groups after the bladder is empty. The primary endpoint is the incidence of urinary dysfunction, which include secondary catheterization or incomplete bladder emptying. Secondary endpoints include urinary tract infection, time to first urination after catheter removal, catheter-related bladder discomfort syndrome, postoperative morbidity and mortality, as well as urinary function within 30 days.

This trial aims to investigate whether ICCAUT strategy, achieved through intermittent clamping of the catheter combined with active urination training in patients undergoing rectal cancer surgery, can impact the rate of urinary dysfunction compared to direct catheter removal. The findings from this study will provide valuable evidence regarding the manipulation of urinary catheters and help guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed preoperative diagnosis of rectal cancer.
2. Patients with tumors located below the rectosigmoid junction (12 cm from the anal verge), as determined by preoperative computed tomography (CT) or rectal magnetic resonance imaging (MRI).
3. Patients undergoing laparoscopic or robotic-assisted total mesorectal excision (TME) for rectal cancer.

Exclusion Criteria:

1. History of abdominal surgery involving the rectum, sigmoid colon, left hemicolectomy, bladder resection or partial resection, prostate surgery, or hysterectomy.
2. History of urethral injury, cranial surgery, spinal surgery, stroke with limb dysfunction, or Parkinson's disease.
3. Inability to urinate through the urethra preoperatively due to various reasons (e.g., ureteral puncture or ureterostomy).
4. Presence of urinary tract infection preoperatively.
5. Previously diagnosed with bladder overactivity syndrome, urinary retention or voiding dysfunction, or diabetic bladder disease.
6. Concomitant resection of other pelvic organs was performed during surgery, including the bladder, prostate, uterus, cervix, and vagina, except for simple adnexal resection.
7. Lateral lymph node dissection for rectal cancer.
8. Injury to the ureter, bladder, or urethra during the perioperative period.
9. Preoperative renal dysfunction (serum creatinine level >133 μmol/L).
10. Emergency surgery.
11. Male patients with preoperative benign prostatic hyperplasia receiving medication treatment.
12. Patients with a ureteral stent or ureteral stricture, or bilateral hydronephrosis.
13. Conversion to open surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Rate of urinary dysfunction | within 7 days after the first time of urethral catheter removal
  Urinary dysfunction is defined as the presence of residual urine volume greater than 100ml, as estimated by bladder ultrasound, after the first voiding following catheter removal, or the need for a second catheterization.

SECONDARY OUTCOMES:
Rate of Urinary tract infections | within 1 days after the first time of urethral catheter removal
  A urinary tract infection is characterized by an inflammatory response in the urinary tract epithelium resulting from bacterial invasion. To diagnose a urinary tract infection, the following criteria must be met simultaneously: 1) urinalysis indicating a bacterial count above the upper limit of normal and 2) positive urine culture.
The time to first voiding after catheter removal | within 1 days after the first time of urethral catheter removal
  The time to first voiding after catheter removal refers to the duration, measured in hours, from the moment the catheter was removed until the patient spontaneously voids for the first time.
Graded assessment of catheter-related bladder discomfort (CRBD) | within 1 days after the first time of urethral catheter removal
  CRBD is a questionnaire given to the patients, to investigate the severity of the discomfort of patients to the urinary catheter
International Consultation on Incontinence Questionnaire-Short Form | on the second day after the first time of urethral catheter removal, and at the 30th day after surgery
  International Consultation on Incontinence Questionnaire-Short Form is used to evaluate the incontinence of voiding. The minimum value is 0 and maximum value is 21. A higher score means a worse outcome
Postoperative complications | within 30 days after the operation
  Complications that occur within 30 days after the operation will be evaluated and documented according to the Clavien-Dindo classification. Complications of grade II or higher were analyzed.
International Prostate Symptom Score | on the second day after the first time of urethral catheter removal, and at the 30th day after surgery
  International Prostate Symptom Score is used to evaluate the severity of urinary difficulties. The scoring range ranges from 0 to 35 points for asymptomatic to severe symptoms. There are three levels of severity: 0-7 is mild, 8-19 is moderate, and 20-35 is severe.
Incidence rate of residual urine volume greater than 200 ml after the first voiding | within 1 days after the first time of urethral catheter removal
  Incidence rate of residual urine volume greater than 200 ml after the first voiding

CONTACTS AND LOCATIONS:
Overall Officials: Yuchen Guo, Ph.D., Principal Investigator — The First Hospital of Jilin University
Locations (2):
- China (2):
  - Firs Hospital of Jilin University, Changchun, Jilin
  - First Hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: Yes
If other researchers can provide valid reasons or demonstrate a need for additional collaboration, we may consider to share the data upon their request after we complete our study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after we complete our study.
Access Criteria: Researchers can provide valid reasons or demonstrate a need for additional collaboration with us.

REFERENCES:
- [Derived] He T, Liang S, Guan Y, Sun J, Hu H, Wang Q, Guo Y. Effect of intermittent urethral catheter clamping combined with active urination training (ICCAUT) strategy on postoperative urinary dysfunction after radical rectal cancer surgery: single-centre randomised controlled trial (ICCAUT -1) study protocol. BMJ Open. 2025 Feb 5;15(2):e095217. doi: 10.1136/bmjopen-2024-095217. PMID 39909516

DOCUMENTS (2):
  • Study Protocol (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT06241703/Prot_003.pdf
  • Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT06241703/SAP_004.pdf